CLINICAL TRIAL: NCT04050800
Title: Characterizing the Safety of [Carbon-11]Butanol and Estimating the Test-Retest Variance in Measurements of Its Whole Body Biokinetics Under Zero-Biological-Change Conditions
Brief Title: Carbon-11 Butanol: Whole Body Radiochemical and Radiation Safety
Acronym: [11C]Butanol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-05020069
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Neuro-Degenerative Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Controls (Experimental): Subjects will be administered two sequential doses of the radiopharmaceutical under nearly zero-biological-change conditions.
  Interventions: Drug: Carbon 11 Butanol

INTERVENTIONS:
Drug: Carbon 11 Butanol — Two sequential administrations of a PET tracer
  Other Names: [11C]Butan-1-Ol

SUMMARY:
This will be a Phase 1, open label, imaging study of radiochemical and radiation safety in healthy volunteers. Using positron emission tomography (PET) and in-line computed tomography (CT), the whole body (WB) biokinetics of Carbon-11 butanol will be quantified with serial scans acquired every 3 minutes for two hours. Vital signs (VS), electrocardiograms (ECGs) and clinical laboratory tests of intrernal organ function will be acquired before and at several timepoints after administration of the radiopharmaceutical. Radiation exposures will be estimated with the MIRD Formalism.

DETAILED DESCRIPTION:
Vital signs (VSs) will be measured, electrocardiograms (ECGs) will be acquired, and blood will be sent to the clinical laboratory for safety assessments before a single dose, intravenous (IV) administration of 555 MBq of Carbon-11 butanol. VSs will be re-measured, ECGs will be acquired again, and more blood will be sent to the clinical laboratory for repeat safety assessments after 2 hours of whole body (WB) scanning. WB scanning will consist of imaging acquisition sweeps of 200 cm from head-to-toe over 180 secs (3 min). Up to 40 sweeps per imaging session will be performed. The subjects will then be given a rest period ("coffee break") for about two hours, after which the entire sequence of events will be repeated. The primary outcome measure will be related to radiation safety derived from the areas under the time-activity curves (AUCs) for internal organs. Co-primary clinical safety measures will include changes in VSs, ECG parameters such as the PR and corrected QT intervals, and clinical laboratory tests, such as proteins that reflect renal and hepatic function. Secondary endpoints will include the time-activity curves (TACs) and total volumes of distribution (VT) in several brain regions. The results should allow calculation of the repeatability coefficients (RCs) under zero-biological-change conditions. RC values will be essential for understanding whether future measurements of effect sizes in response to therapeutic maneuvers or the differences between groups are meaningful.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent.
* age 18-89
* Subjectively healthy and, in the opinion of the investigators, likely to tolerate the imaging procedures and be compliant with the schedule of follow up telephone calls.
* Normal hemodynamic function. Systolic blood pressure and pulse must be higher than 120 mmHg and 60 beats per minute while sitting. At the discretion of the investigators, people who regularly engage in vigorous exercise more than four times per week may be enrolled if their systolic blood pressure and pulse are higher than 100 mmHg and 50 beats per minute while sitting.
* Unremarkable electrocardiograms, with PR intervals of less than 200 mSec and QTcF intervals (corrected with Frederica's method) of less than 440 mSec.
* No concurrent medications with the exception of p.r.n. NSAIDS, which must be discontinued one week prior to PET scanning.
* Willing and able to refrain from abusing any recreational drugs, including marijuana, and drink less than one unit of alcoholic beverages per day starting one week prior to PET scanning, and avoided for the next four weeks.
* Willing to refrain from donating blood for four (4) weeks before the study and for four (4) weeks after the study.
* Willing to refrain from participating in any other research study that requires taking medication for four (4) weeks before the study and for four (4) weeks after the study.
* Willing to refrain from being vaccinated for four (4) weeks before the study and for four (4) weeks after the study.
* All clinical laboratory test results within normal limits or not clinically significant. For example, elevated bilirubin levels in subjects with Gilbert's syndrome will be allowed, as will small red blood cell volumes in healthy people with sickle cell trait.

Exclusion Criteria:

* Subjects may not be a member of a vulnerable population.
* Women may not be pregnant or breast feeding.
* History of multiple hypersensitivity reactions (atopia), as indicated by allergies to multiple medications, foods, and seasonal pollens.
* History, physical examination, or clinical laboratory tests suggestive of a condition, disorder, or disease that could adversely affect drug absorption, distribution, metabolism, or elimination (ADME) of the tracer, including chronic liver or renal failure.
* Positive urine toxicology screen for recreational drugs other than marijuana.
* May not have taken any controlled medications, including other study drugs, in the 30 days prior to PET scanning or for 10 half-lives, whichever is longer.
* May not have donated blood in the 30 days prior to PET scanning.
* May not have participated in research administering drugs in the last 30 days.
* May not have been vaccinated in the 30 days prior to PET scanning.
* May not have been exposed to radiation during research of more than 10 mSv during the last year.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Effective Dose (ED) | Day 1, from the measurements of exposures during the first 2 hours post administration.
  Fundamental radiation dose quantity in the International Commission on Radiological Protection (ICRP) system of radiological protection. Calculated with OLINDA-EXM software (OLINDA/EXM stands for Organ Level INternal Dose Assessment/EXponential Modeling).

SECONDARY OUTCOMES:
Change in Radiochemical Safety Assessments | Pulse at two hours post administration compared to pulse shortly before administration.
  Change in pulse
Change in Radiochemical Safety Assessments | Blood pressure at two hours post administration compared to blood pressure shortly before administration.
  Change in blood pressure
Change in Radiochemical Safety Assessments | At two hours post administration compared to same parameters shortly before administration.
  Change in heart rhythm on electrocardiogram (ECG)
Change in number of Subjects with prolonged PR interval greater than 20 mSec | At two hours post administration compared to same parameters shortly before administration.
  Change in PR interval on electrocardiogram (ECG)
Change in number of subjects with QTc >440 mSec | At two hours post administration compared to same parameters shortly before administration.
  Change in corrected QT interval on electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Overall Officials: P. David Mozley, MD, Principal Investigator — Cornell University Weill College of Medicine
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be shared. The investigators will attempt to contribute the "raw" imaging data to a public archive for curation.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon publication of the results.
Access Criteria: Any investigators with a reasonable request for the data.